CLINICAL TRIAL: NCT00798577
Title: Study of the Progression of Bacterial Conjunctivitis Symptoms Upon Antibiotic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Topical Solutions Ltd. (Industry)
Responsible Party: Paul Cockrum, PhD, Director - Medical Affairs, Alcon Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMA-08-03
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Bacterial Conjunctivitis
Keywords: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vigamox (Experimental): Vigamox Ophthalmic Solution (Moxifloxacin 5mg/mL)
  Interventions: Drug: Vigamox Ophthalmic Solution
- BSS Placebo (Placebo Comparator): Balanced Salt Solution
  Interventions: Drug: BSS placebo

INTERVENTIONS:
Drug: Vigamox Ophthalmic Solution — Moxifloxacin 5mg/mL 3 times daily for 7 days
  Arms: Vigamox
Drug: BSS placebo — Balanced Saline Solution for 3 doses, then Moxifloxacin 5mg/mL 3 times daily for 7 days
  Arms: BSS Placebo

SUMMARY:
The primary objective of this study is to investigate the initial antibiotic effects in the treatment of bacterial conjunctivitis symptoms in subjects one year of age and older.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis in one or both eyes of bacterial conjunctivitis based on:

   * symptoms less than or equal to 24 hours prior to first visit
   * rating > or equal to 1 for bulbar conjunctival injection
   * must have a rating > 1 for conjunctival discharge / exudate in at least one eye (the same eye as bulbar conjunctival injection ) at Visit 1, and
2. Must experience some matting in the affected eye(s).
3. 1 year of age or older, of any race and either sex
4. Able to understand and sign an informed consent that has been approved by an Institutional Review Board; or if the subject is a minor, the informed consent must be signed and understood by the subjects legally authorized representative (parent or guardian). Assent to participate should be obtained from subjects 6 years of age or older unless not allowed by local regulation.
5. Must agree to comply with study visit schedule, photographs and other study requirements. If subject is a minor, the parent or guardian must agree to ensure compliance.

Exclusion Criteria:

1. Cannot have had bacterial conjunctivitis as reported by subject (or parent if subject is a minor) for > 24 hours.
2. Any current lid disease on clinical examination.
3. Known or suspected allergy or hypersensitivity to fluoroquinolones.
4. Suspected fungal, viral (e.g. Herpes simplex) or Acanthamoeba infection, based on clinical observation.
5. Any systemic or ocular disease or disorder, complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study (e.g., hepatitis, acute or chronic renal insufficiency).
6. Use of topical ocular medications during the study period.
7. Antibiotics (systemic or topical) may not be used within 7 day of visit 1 or anytime after this visit for the duration of the study.
8. Women of childbearing potential not using reliable means of birth control.
9. Women who are pregnant or lactating.
10. Enrollment of more than one person per household at the same time.
11. Enrollment of the investigator or his or her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of these individuals.
12. Participation in any investigational drug or device study within 30 days of entering this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vigamox: Vigamox Ophthalmic Solution (Moxifloxacin 5 mg/mL) three times daily for 7 days
- Placebo: Balanced Salt Solution (BSS) placebo for 3 doses, then Moxifloxacin 5mg/mL 3 times daily for 7 days
Period: Overall Study
Arm/Group | Vigamox | Placebo
Started | 17 | 7
Completed | 17 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vigamox | Placebo | Total
Number analyzed (Participants) | 17 | 7 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 7 | 14
  Between 18 and 65 years | 10 | 0 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Exploratory Outcomes From Digital Photography
Description: Photographs were taken before and after treatment. Outcome is the number of patients whose photographs showed a subjective visual change based upon an exploratory review of patient photographs in signs of bacterial conjunctivitis before and after treatment.
Time Frame: 24 hours after administration of first dose
Measure: Number; unit: Participants
Arm/Group | Vigamox | Placebo
Number analyzed (Participants) | 17 | 7
Participants | 17 | 7

2. Secondary Outcome: Exploratory Evaluation of Changes in Ocular Signs and Symptoms
Description: Number of patients who had clinical resolution (0 on all scales below) from baseline (Day 1) to Day 2 in ocular and symptoms of bacterial conjunctivitis:
  Bulbar Conjunctival Injection - 0 (none) to 4 (Severe) scale. Conjunctival Discharge (Mucopurulent) - 0 (none) to 3 (Severe) scale. Lid Erythema - 0 (none) to 3 (Severe) scale. Lid Swelling - 0 (none) to 3 (Severe) scale. Palpebral Conjunctiva - 0 (none) to 3 (Severe) scale. Foreign Body Sensation - 0 (none) to 3 (Severe) scale. Tearing - 0 (none) to 3 (Severe) scale. Photophobia - 0 (none) to 3 (Severe) scale.
Time Frame: Baseline (Day 1) to Day 2
Measure: Number; unit: Participants
Arm/Group | Vigamox | Placebo
Number analyzed (Participants) | 17 | 7
Participants | 17 | 7

3. Secondary Outcome: Microbiological Culture Evaluation/Eradication Percent - Enterobacter Faecalis and Candida Albicans
Description: Eradication percent (absence of specified bacteria) of each bacteria identified at Day 1
Time Frame: 24 hours after administration of first dose
Measure: Number; unit: Percent bacteria eradicated
Arm/Group | Vigamox | Placebo
Number analyzed (Participants) | 17 | 7
Percent bacteria eradicated
  Enterobacter faecalis | 17 | 100
  Candida albicans | 75 | 0

4. Secondary Outcome: Microbiological Culture Evaluation/Eradication Percent - Eradication of All Other Isolates and Corynform-like
Description: Eradication percent (absence of specified bacteria) of each bacteria identified at Day 1
Time Frame: 24 hour after administration of first dose
Population: No patients in the Placebo group had Corynform-like bacteria (or other types of bacteria) identified at Day 1
Measure: Number; unit: Percent bacteria eradicated
Arm/Group | Vigamox | Placebo
Number analyzed (Participants) | 17 | 0
Percent bacteria eradicated
  Eradication of all other isolates | 100 |
  Corynform-like | 0 |

5. Secondary Outcome: Microbiological Culture Evaluation/Eradication Percent - Staphylococcus Aureus, Steptococcus Pneumoniae, and Enterobacter Cloacae
Description: Eradication percent (absence of specified bacteria) of each bacteria identified at Day 1
Time Frame: 24 hours after administration of first dose
Population: No patients in the Vigamox group had Staphylococcus aureus, Steptococcus pneumoniae, or Enterobacter cloacae identified at Day 1.
Measure: Number; unit: Percent bacteria eradicated
Arm/Group | Vigamox | Placebo
Number analyzed (Participants) | 0 | 7
Percent bacteria eradicated
  Staphylococcus Aureus |  | 0
  Steptococcus Pneumoniae |  | 50
  Enterobacter Cloacae |  | 67

ADVERSE EVENTS:
Arm/Group | Vigamox | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/7
Other Adverse Events (participants affected / at risk) | 0/17 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All presentations/publications of study results are subject to Alcon approval.